CLINICAL TRIAL: NCT05426915
Title: Clinical Study for the Effectiveness of Roflumilast Treatment in COPD Greek Patients Based on Standard Clinical Practice. An Observational, Non-interventional Multicenter Study.
Brief Title: Clinical Study for the Effectiveness of Roflumilast Treatment in COPD Greek Patients Based on Standard Clinical Practice.
Acronym: ARGO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-ROFDAM-EL-161
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Copd; COPD Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preferred pharmacological management for COPD according to the GOLD guidelines are the long-acting anticholinergic LAMAs (Long-Acting / Short-Acting Muscarinic Antagonists), and long-acting β 2-Agonists LABA (Long-acting LABA) / β2-Long Action Fighters) as well as inhaled corticosteroids (ICS) Other drugs that can be used besides long-acting, are short-acting anticholinergics (SAMA) and β2-agonists (SABA), methylxanthines (Aminophylline and Theophylline), mucolytics and phosphodiesterase inhibitors 4 (Phosphorus) of which is roflumilast

DETAILED DESCRIPTION:
Roflumilast is a phosphodiesterase 4 (PDE4) inhibitor, a non-steroidal, anti-inflammatory active substance intended to target both systemic inflammation and COPD-related lung inflammation. The mechanism of action is the inhibition of PDE4, which is an important enzyme for the metabolism of cyclic adenosine monophosphate (cAMP) found in structural and inflammatory cells, which are important in the pathogenesis of COPD. Roflumilast targets PDE4A, 4B and 4D subtypes with similar activity in the nanomolecular range. The affinity for PDE4C subtypes is 5 to 10 times lower. This mechanism of action and selectivity also apply to roflumilast N-oxide, which is the main active metabolite of roflumilast. Inhibition of PDE4 leads to increased levels of intracellular cAMP and attenuates COPD-related dysfunctions of leukocytes, smooth muscle cells of the airways and lungs, endothelial cells and epithelial cells and epithelial cells. In vitro stimulation of human neutrophils, monocytes, macrophages or lymphocytes, roflumilast and roflumilast N-oxide suppress the release of inflammatory mediators e.g. leukotriene B4, reactive oxygen species, tumor necrosis factor α, interferon γ and granzyme B.

In patients with COPD, roflumilast reduced neutrophils in the sputum. In addition, it mitigated the influx of neutrophils and eosinophils into the airways of healthy volunteers following endotoxin challenge. Studies using roflumilast have shown that there has been a statistically significant and clinically significant reduction in exacerbations in COPD patients. Depending on the study, a reduction ranging from 15% -37% was observed. In 2 placebo-controlled 12-month roflumilast studies, where 50% of patients were on maintenance therapy with a LABA, the reduction in exacerbations was 17% (P <0.001) (12). Also, in 2 studies of roflumilast for 6 months, controlled with placebo, the reduction of exacerbations when taken with salmeterol was 37%, P = 0.0315 (post-hoc analysis) or with Tiotropium 23%, P = 0.196.

The drug of the present study is Damirast 500 mg of which the active substance is roflumilast. It is a potent selective PDE4 inhibitor with multiple anti-inflammatory actions. Improves pulmonary function (48-55mL), reduces exacerbations (15-37%)and prolongs the time to the first exacerbation (up to 40%).

Damirast is indicated for the maintenance treatment of severe chronic obstructive pulmonary disease (COPD) in addition to bronchodilator therapy, LABA / LAMA and / or inhaled corticosteroids.

Damirast is an innovative anti-inflammatory treatment specifically designed for COPD patients with chronic cough and sputum. The anti-inflammatory action of Damirast reduces the incidence of exacerbations, while it also actively contributes to the improvement of the patient's lung function, making it the appropriate medication for the long-term treatment of COPD. In addition, once daily oral administration is expected to play a key role in patient compliance, as it offers the added benefit of systematic availability and easy access. Damirast can thus reach even the smallest and most distant bronchi and pulmonary alveoli, which are often blocked by mucus, making it difficult to exchange gases and prevent the absorption of inhaled drugs.

ELIGIBILITY:
Inclusion criteria

1. Adult patients indicated for maintenance treatment of severe COPD associated with chronic bronchitis with a history of frequent exacerbations in addition to bronchodilator / ICS therapy.
2. Consent and compliance with the therapies and study procedures. Exclusion criteria According to the contraindications of the SPC of the product. Patients should not take theophylline.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with COPD which is now one of the top three causes of death worldwide. In Greece there are about 700,000 patients with COPD (prevalence 10.6%) and similar is the global prevalence (9-10%) of the disease for adults over 40 years.
  Preferred pharmacological management for COPD according to the GOLD guidelines are the long-acting anticholinergic LAMAs (Long-Acting / Short-Acting Muscarinic Antagonists), and long-acting β 2-Agonists LABA (Long-acting LABA) / β2-Long Action Fighters) as well as inhaled corticosteroids (ICS).
  Other drugs that can be used besides long-acting, are short-acting anticholinergics (SAMA) and β2-agonists (SABA), methylxanthines (Aminophylline and Theophylline), mucolytics and phosphodiesterase inhibitors 4 (Phosphorus) of which is roflumilast.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
change in CCQ | 12 months
  (Clinical COPD Questionnaire) changes in 3-6-9-12 months

SECONDARY OUTCOMES:
change in mMRC | 12 months
  (Modified Medical Research Council) changes in 3-6-9-12 months
change in CAT | 12 months
  (COPD Assessment Test) changes in 3-6-9-12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sotiria Hospital, Athens, Attica, Greece